CLINICAL TRIAL: NCT06209216
Title: An Observational Study to Explore Twenty-Four Seven Functional Status Measures in Total Hip Replacement (LEARNT)
Brief Title: Twenty-Four Seven Functional Status in Total Hip Replacement
Acronym: LEARNT
Status: Completed | Type: Observational
Sponsor: Koneksa Health (Industry)
Responsible Party: Sponsor
Other Study IDs: KH009
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Total Hip Replacement
Keywords: Functional Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Hip Replacement: No intervention

SUMMARY:
The goal of this observational study is to define digital remote monitoring measures for functional status (activities of daily living) in patients receiving total hip replacement. Functional status will be collected using a study iPhone and two wearable wrist monitors.

DETAILED DESCRIPTION:
Approximately 25 participants will be enrolled in this study. The study consists of a 1-week Screening period, a 1-week Baseline period, up to 6-week assessment period (post-surgery), and an end of participation (EOP) visit. With the exception of in clinic visits at the beginning and end of study, this observational study will leverage fully remote data capture.

The categories of functional status and corresponding measures captured in this study include:

1. Physical activity and mobility, with outcome measures including hourly and daily step count, gait speed, and metabolic equivalent of task.
2. Vital signs, with outcome measures including heart rate, heart rate variability and blood pressure.
3. Sleep concept, with outcome measures including sleep duration, sleep quality, sleepiness and sleep timing.
4. HRQoL captured using validated instruments and diaries via electronic patient reported outcomes (ePRO) platforms, assessing aspects of health that are meaningful to individual's hip replacement such as disease- and treatment-related symptoms and the impact their physical health may have on activities of daily living, their work life, and socializing.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with osteoarthritis of the hip or degenerative joint disease and have decided to undergo total hip arthroplasty
2. Patients willing to sign the informed consent form
3. Age 30 and older
4. Demonstrated ability to perform satisfactory at-home assessments as well as the mobile application to synchronize data collection and respond to questionnaires during the screening period

Exclusion Criteria:

1. Participants with clinically unstable serious diseases (e.g., heart or lung disease) that would deem them unfit for the study in the Investigator's opinion
2. Secondary total hip replacement on the same side
3. Hip replacement for neoplasm, proximal femoral fracture, or other causes than osteoarthritis
4. Contemporary bilateral replacement
5. History of substance abuse in the last 6 months, excluding medical or recreational non-inhaled marijuana
6. Current cancer
7. Presence of neurological diseases previous to and/or following surgery (peripheral neuropathy is generally acceptable)
8. Congenital abnormalities
9. Patients with active infection within last 30 days
10. Psychotropic drugs except for pain management and antidepressants

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants requiring total hip replacement surgery will participate in this study for ~6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Overall Hip Assessment - In Clinic | Baseline Day 1 through Day 42 End of Participation
  Harris Hip Score
Mobile Vital Signs via Mobile Blood Pressure Cuff | Baseline Day 1 through Day 42 End of Participation
  Orthostatic blood pressure
Daily Measurements via Wrist-worn Device | Baseline Day 1 through Day 42 End of Participation
  Heart rate variability, body temperature, step count, blood oxygen saturation
Objective Measures of Sleep via Wrist-worn Device | Baseline Day 1 through Day 42 End of Participation
  Sleep staging measured by a combination of heart rate variability + actigraphy + blood oxygen saturation and vital signs during sleep
Motor Function Assessments via Koneksa Application | Baseline Day 1 through Day 42 End of Participation
  Gait (20 second walk test)
Participant Diary via Koneksa Application | Baseline Day 1 through Day 42 End of Participation
  Pain level likert scale, pain medication use, walking aid use
Sleep Electronic Patient Reported Outcomes | Baseline Day 1 through Day 42 End of Participation
  Sleep Diary and Stanford Sleepiness Scale
Quality of Life Patient Reported Questionnaire Scores | Baseline Day 1 through Day 42 End of Participation
  Instrumental Activities of Daily Living Scale, PHQ-9 for Depression Score, Functional Assessment of Chronic Illness Therapy - Fatigue (PROMIS SF v1.0 Fatigue 13a) Score, Brief Pain Inventory Short Form for Pain Score
Additional Questionnaire via Koneksa Platform | Baseline Day 1 through Day 365 End of Participation
  Usability for devices and app-based study-specific assessments questionnaire, questionnaires for site clinical care team likelihood to recommend all devices used, and app-based assessments, questionnaires for understanding of tasks and assessment of meaningfulness, participant and/or caregiver likelihood to recommend, ease of use and satisfaction
Clinician Reported Adverse Events | Baseline Day 1 through Day 365 End of Participation
  Clinical event defined as event requiring medical intervention from call to doctor or emergency room services (such as fall)

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Medical Associates, The Villages, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided